CLINICAL TRIAL: NCT04851834
Title: A Phase 1/2, Open-label, Dose-exploration and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NTX-301 Monotherapy in Advanced Solid Tumours, and in Combination With Platinum-based Chemotherapy in Advanced Ovarian & Bladder Cancer, and in Combination With Temozolomide as Adjuvant (Maintenance) Therapy in High-grade Glioma (Optional Arm)
Brief Title: NTX-301 Monotherapy in Advanced Solid Tumours and in Combination With Platinum-based Chemotherapy in Advanced Ovarian & Bladder Cancer and in Combination With Temozolomide in High-grade Glioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated by IP Holder (collaborator), PinotBio Inc.
Sponsor: Xennials Therapeutics Australia Pty Ltd (Industry)
Collaborators: Pinotbio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XNTR-20-02
Record Dates: First submitted 2021-04-08; First posted 2021-04-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumor; Platinum-Resistant Ovarian Cancer; Platinum-Resistant Urothelial Carcinoma; High-grade Glioma
Keywords: Hypomethylating Agent; Nucleoside Analog; DNA Demethylation; Solid Tumors; Ovarian Neoplasms; Urinary Bladder Neoplasms; Platinum-resistant; Carboplatin; Cisplatin; Glioma; IDH1; Temozolomide
MeSH Terms: conditions — Glioma; Ovarian Neoplasms; Urinary Bladder Neoplasms | interventions — Platinum Compounds; Cisplatin; Carboplatin; Temozolomide

STUDY DESIGN:
Intervention Model Description: Dose escalation to determine MTD/RP2D, then dose expansion
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- NTX-301 Monotherapy Dose Escalation (Experimental): NTX-301 monotherapy dose escalation in patients with advanced solid tumours
  Interventions: Drug: NTX-301
- NTX-301 platinum-based doublet therapy Dose Escalation (Experimental): NTX-301 combined with platinum-based chemotherapy in platinum-resistant advanced ovarian & bladder cancer
  Interventions: Drug: NTX-301; Drug: Platinum-based Chemotherapy
- NTX-301 platinum-based doublet therapy Dose Expansion (Experimental): NTX-301 combined with platinum-based chemotherapy in platinum-resistant advanced ovarian & bladder cancer
  Interventions: Drug: NTX-301; Drug: Platinum-based Chemotherapy
- NTX-301 Temozolomide doublet therapy Dose Escalation (Experimental): NTX-301 combined with Temozolomide (TMZ) as adjuvant (maintenance) treatment in IDH1 mutated high-grade glioma
  Interventions: Drug: NTX-301; Drug: Temozolomide
- NTX-301 Temozolomide doublet therapy Dose Expansion (Experimental): NTX-301 combined with Temozolomide (TMZ) as adjuvant (maintenance) treatment in IDH1 mutated high-grade glioma
  Interventions: Drug: NTX-301; Drug: Temozolomide

INTERVENTIONS:
Drug: NTX-301 — Oral hypomethylating agent
Drug: Platinum-based Chemotherapy — Standard of care for ovarian and bladder cancer
  Other Names: Cisplatin; Carboplatin
  Arms: NTX-301 platinum-based doublet therapy Dose Escalation; NTX-301 platinum-based doublet therapy Dose Expansion
Drug: Temozolomide — Standard of care for high-grade glioma
  Arms: NTX-301 Temozolomide doublet therapy Dose Escalation; NTX-301 Temozolomide doublet therapy Dose Expansion

SUMMARY:
This is a Phase 1/2, open-label, dose-exploration, combination/expansion study, which will start by evaluating the safety and tolerability of NTX-301, an oral DNMT1 inhibitor, as a monotherapy in patients with advanced solid tumours, who have failed treatment with available therapies known to be active for treatment of their corresponding disease. It will then explore the safety and tolerability of NTX-301 in combination with platinum-based therapy in patients with ovarian and bladder cancer. Optionally, the safety and tolerability of NTX-301 in combination with Temozolomide (TMZ) in patients with Isocitrate Dehydrogenase 1 (IDH1) mutated high-grade glioma will also be assessed.

DETAILED DESCRIPTION:
Dose Exploration (Phase 1a, n~25): This part of the study will assess the safety and tolerability of NTX-301 and to identify the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D). It will initiate with a dose escalation using a 3+3 design.

Combination Dose and Disease Expansion (Phase 1b-2a, n~60): The study will be expanded in specific subsets of patients with solid tumours and with combination therapy as follows:

* Arm 1 (Phase 1b, n~20): Dose Escalation, NTX-301 platinum-based doublet therapy
* Arm 2 (Phase 2a, n~40): Dose Expansion, NTX-301 platinum-based doublet therapy

Patients with advanced ovarian & bladder cancer considered to be incurable by the investigator and for which available anti-cancer therapy has been exhausted will be enrolled for this component. Patients will be given NTX-301 at the MTD determined in Phase 1a. This will be combined with a platinum-based agent that will be administered by IV infusion.

Optional Cohort -High-Grade Glioma Combination Dose & Disease Expansion (Phase 1b-2a, n~40)

* Arm 3 (Phase 1b, n~20): Dose Escalation, NTX-301 combination therapy with TMZ
* Arm 4 (Phase 2a, n~20): Dose Expansion, NTX-301 combination therapy with TMZ

Patients with IDH1 mutated high-grade glioma that have commenced initial chemoradiotherapy with temozolomide and are yet to commence Temozolomide maintenance therapy will be enrolled for this component. Patients will be given NTX-301 at the MTD determined in Phase 1a. This will be combined with TMZ that will be administered orally.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and be willing to sign an informed consent form.
2. Male or female, ≥ 18 years old at the time of screening.
3. Diagnosis of histologically or cytologically confirmed:

   1. Locally advanced or metastatic cancer (all solid tumours). Subjects must be considered refractory or intolerant to SOC therapies or have refused standard therapy. If the last treatment a subject received was an inhibitor of DNA synthesis or a hypomethylating agent, at least 5 half-lives must have passed prior to commencing treatment. (Phase 1a, Dose Escalation Monotherapy), OR
   2. Locally advanced or metastatic cancer (ovarian or bladder cancer and other solid tumours where in the opinion of the investigator, retreatment with cisplatin or carboplatin may be beneficial to the subject). Subjects must be considered refractory or intolerant to SOC therapies or have refused standard therapy, in such a case, reason for the refusal to be captured in Case Report Form (CRF). If subject is having a drug holiday to recover from cisplatin toxicity, entry to the trial is allowed if the PI feels the subject will receive further benefit from cisplatin, the toxicity has recovered to ≤ CTCAE Grade 1 and all other eligibility criteria are met. Last treatment prior to trial entry with a platinum is not required. If the last treatment a subject received was an inhibitor of DNA synthesis or a hypomethylating agent, at least 5 half-lives must have passed prior to commencing study treatment). (Phase 1b, Dose & Disease Expansion Combination Arms, Arms 1 & 2), OR
   3. High-grade glioma, such as glioblastoma multiforme (GBM) that are:

   Newly diagnosed and are undergoing, or are planned to undergo, 42 Days of SOC chemoradiation therapy as per part 1 of the eviQ protocol 3364 v.1. Subjects successfully enrolled will receive a subsequent combination of NTX-301, Days 1-5 and 8-12 as well Temozolomide on Days 15-19 of their first 28-Day cycle of part 2 of the eviQ protocol 3364 v.1. This combination arm replaces the Temozolomide monotherapy SOC maintenance therapy as described in Part 2 of the eviQ protocol 3364 v.1. In order to prevent any potential delays after radiotherapy, subjects can be enrolled at any time during Chemoradiation (eviQ Part 1). In order to commence the TMZ combination arms the subject is required to complete the full 42 Days of eviQ part 1, and also receive their first dose of the TMZ combination arm within the screening window. This timing can be adjusted based on medical need on a subject-by-subject basis as per the discretion of the principal investigator together with the approval of the medical monitor (Phase 1b, 2a, Dose & Disease Expansion Combination GBM (optional) Arm, Arms 3 & 4) Note: subjects must also have at least one measurable disease lesion per RECIST 1.1 &/or RANO criteria. For Phase 1a only, non-measurable disease may also be included based on PI and MM discretion on a case-by-case basis.
4. Eastern Cooperative Oncology Group performance status of 0 to 1
5. Able to take oral medications and willing to record daily adherence to the study drug.
6. Cardiac

   1. QT interval corrected using the Fridericia method (QTcF) ≤ 450 msec for males and ≤ 470 msec for females at screening and on Day 1, prior to dose administration (the mean of triplicate measurements will be used to determine eligibility)
   2. LVEF >45% based on ECHO Scan within 60 Days of screening.
7. Evidence of adequate hepatic function at screening, as defined by the following:

   1. AST and ALT ≤2.5 × upper limit of normal (ULN) (≤5 × ULN if liver metastases are present); and
   2. Total bilirubin ≤1.5 × ULN (< 2.0 x ULN for subjects with liver metastases or documented Gilbert's syndrome).
8. Adequate haematology laboratory assessment at screening, as defined by:

   1. Absolute neutrophil count ≥1.00 x109/L;
   2. Haemoglobin ≥90 g/L; and
   3. Platelet count ≥100 x109/L.
9. Evidence of adequate renal function, as defined by a calculated creatinine clearance ≥45 mL/min using the Cockcroft-Gault equation, renal nuclear medical scan, or a 24-hour urine collection with plasma and urine creatinine concentrations respectively. There can be exceptions on a case-by-case basis as per the discretion of the principal investigator and approval by the Medical Monitor and Sponsor.
10. Adequate coagulation laboratory assessments (i.e., within normal reference range values) at screening, in the opinion of the Investigator.
11. Female subjects must:

    1. Be of non-child-bearing potential i.e. surgically sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before the Screening visit) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone level consistent with postmenopausal status, per local laboratory guidelines), or
    2. If of child-bearing potential, must agree not to attempt to become pregnant, must not donate ova, and, if engaging in sexual intercourse with a male partner, must agree to use an acceptable method(s) of contraception from signing the consent form until at least 45 Days after the last dose of study drug.
12. Male subjects must agree not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use an acceptable method of contraception from signing the consent form until at least 90 Days after the last dose of study drug
13. Estimated life expectancy of at least 3 months, in the opinion of the Investigator.

    Willing and able to comply with all scheduled visits, treatment plans, laboratory tests, and other study procedures.
14. Willing and able to comply with all scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Investigational agents, including hypomethylating agents, in the past 5 half-lives
2. Patients with symptomatic brain metastases.
3. Evidence of abnormal cardiac function as defined by any of the following:

   1. Myocardial infarction within 6 months of Cycle 1, Day 1
   2. Symptomatic congestive heart failure (New York Heart Association > class II)
   3. Unstable angina
   4. Unstable cardiac arrhythmia. Stable cardiac arrhythmia that is Medically managed is allowable. Borderline subjects are allowable on a case-by-case basis as per the discretion of the Principal Investigator and approval by the Medical Monitor and Sponsor.
4. Unable to swallow oral medications.
5. Gastrointestinal (GI) Gastrointestinal conditions that, in the opinion of the Investigator, could affect the absorption of NTX-301
6. History of bowel obstruction, abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months of the first administration of NTX-301 (Cycle 1, Day 1) (unless otherwise approved by the Investigator).
7. Unless approved by treating physician, use of any herbal or prescription medications, or consumption of foods known to be strong inhibitors of cytochrome P450 3A (CYP3A) enzymes within 7 Days prior to the first administration of NTX-301 (Cycle 1, Day 1). These include (but are not limited to):

   1. Certain Medications defined within the study protocol
   2. Foods: Grapefruit or Seville orange (or grapefruit- or Seville orange-containing products, including juices).
8. Use of any herbal or prescription medications known to be strong inducers of CYP3A enzymes within 7 Days prior to the first administration of NTX-301 (Cycle 1, Day 1)
9. Clinically significant active infection within 2 weeks of the first dose of NTX-301 (Cycle 1, Day 1).
10. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at the Screening visit.
11. History of other malignancy within the past 2 years, with the following exceptions:

    1. Malignancy treated with curative intent and with no known active disease present for ≥ 2 years before enrolment and felt to be at low risk for recurrence by the treating physician.
    2. Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease.
    3. Adequately treated cervical carcinoma in situ without evidence of disease.
    4. Adequately treated breast ductal carcinoma in situ without evidence of disease.
    5. Prostatic intraepithelial neoplasia without evidence of prostate cancer.
    6. Adequately treated urothelial papillary non-invasive carcinoma or carcinoma in situ.
12. Major surgery within 28 Days of Cycle 1, Day1, with the following exceptions:

    1. Major surgical procedures ≤28 Days of beginning study drug, or
    2. Minor surgical procedures ≤7 Days.
    3. No waiting required following port-a-cath placement or for venous access.
    4. Planned elective surgery unrelated to the subject's oncologic diagnosis, such as hernia repair, may be allowed, at the discretion of the Investigator, as long as it was performed at least 2 weeks prior to starting NTX-301, and the subject has recovered fully from this procedure.
13. Received cancer-directed therapy within the following timeframes:

    1. Anti-tumour therapy (chemotherapy, antibody therapy, molecular targeted therapy, hormonal therapy or investigational agent) within 28 Days or (unless 5 times the half-life is shorter than 28 Days); Note: concurrent use of hormone deprivation therapy for hormone-refractory prostate cancer, bisphosphonate or denosumab for skeletal related events per institution guideline is permitted.
    2. Wide field radiation administered ≤28 Days or limited field radiation for palliation ≤7 Days prior to starting study drug or has not recovered from side effects of radiation therapy.
    3. Receiving treatment with any other concurrent investigational device(s) or conventional agent(s) within 28 Days (unless 5 times the half-life is shorter than 28 Days) of Cycle 1, Day 1.
14. Adverse Events due to investigational or conventional agents >4 weeks earlier that have not recovered to a severity of Grade 0 or Grade 1 (per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 or higher), with the exception of alopecia.

    Note: (applies to Phase 1a, dose levels 3-5 and Phase 1b only):

    i. Subjects with chronic Grade 2 toxicities may be eligible per discretion of the Investigator and Sponsor (e.g., Grade 2 chemotherapy induced neuropathy).

    ii. Grade 2 or 3 toxicities from prior anti-tumour therapy that are considered irreversible - defined as having been present and stable for > 6 months (such as ifosfamide-related proteinuria) may be allowed if they are not otherwise described in the exclusion criteria AND there is agreement to allow by both the Investigator and Sponsor
15. For women of childbearing potential, a positive pregnancy test at screening, or on Day 1, prior to dose administration.
16. Pregnant or breast-feeding (or planning to breastfeed while on study through 15 Days after the last dose of study drug.
17. Hypersensitivity or other clinically significant reaction to the study drug or its inactive ingredients.
18. Known substance abuse or medical, psychological, or social conditions that, in the opinion of the Investigator, may interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
19. Any other condition or prior therapy that in the opinion of the Investigator would make the subject unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements
20. COVID-19 vaccinations: Administration of an approved COVID-19 vaccine less than14 Days prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Safety & Tolerability: Incidence, type, and severity of Adverse Events (AE) | 15 Months
Safety & Tolerability: Dose-limiting Toxicities (DLT) | 15 Months

SECONDARY OUTCOMES:
Incidence of DLTs according to the MTD/RP2D evaluation process | 12 Months
Pharmacokinetics (PK): Maximum observed concentration (Cmax) | 12 Months
Pharmacokinetics (PK): Time to Cmax (Tmax) | 12 Months
Pharmacokinetics (PK): Trough concentrations | 12 Months
Pharmacokinetics (PK): Area under the concentration-time curve (AUC0-t) | 12 Months
Pharmacokinetics (PK): Apparent terminal elimination half-life (t1/2) | 12 Months

OTHER OUTCOMES:
Tumour Response Assessment per RECIST 1.1 &/or RANO criteria | Up to 32 Months
Efficacy: Objective response rate (ORR) | Up to 32 Months
Efficacy: Disease control rate (DCR) | Up to 32 Months
Efficacy: Time to response (TTR) | Up to 32 Months
Efficacy: Duration of response (DOR) | Up to 32 Months
Efficacy: Progression free survival (PFS) | Up to 32 Months
Pharmacodynamics (PD): DNMT1 level | Up to 32 Months
Pharmacodynamics (PD): Global DNA Methylation | Up to 32 Months

CONTACTS AND LOCATIONS:
Overall Officials: Joyce L. Steinberg, MD, Study Director — Xennials Therapeutics Inc
Locations (2):
- Australia (2):
  - St. Vincent's Hospital - The Kinghorn Cancer Center, Darlinghurst, New South Wales
  - St. George Private Hospital, Kogarah, New South Wales